CLINICAL TRIAL: NCT05780086
Title: A Phase I Study to Evaluate the Short-term Safety of and Tolerability to a Sodium-free Peritoneal Dialysis Solution With 30% Icodextrin and 10% Dextrose in Patients in Peritoneal Dialysis, on a Preliminary Basis
Brief Title: Safety of and Tolerability to a Sodium-free Peritoneal Dialysis Solution
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Sequana Medical N.V. (Industry)
Responsible Party: Principal Investigator, Eduardo Almeida Gutiérrez, Head of Research and Education at Hospital de Cardiologia, Instituto Mexicano del Seguro Social
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2022-785-034
Record Dates: First submitted 2023-02-07; First posted 2023-03-22 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Icodextrin; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30% icodextrin and 10% dextrose (Experimental): Dwell time of 24 hours using a 500 ml sodium-free peritoneal dialysis solution based on 30% icodextrin and 10% dextrose
  Interventions: Drug: 30% icodextrin and 10% dextrose

INTERVENTIONS:
Drug: 30% icodextrin and 10% dextrose — Dwell time of 24 hours using a 500 ml sodium-free peritoneal dialysis solution based on 30% icodextrin and 10% dextrose

SUMMARY:
This study will evaluate the safety and tolerability profile of a dwell time (bath) of 24 hours using a 500 ml sodium-free peritoneal dialysis solution based on 30% icodextrin and 10% dextrose in patients with chronic kidney failure undergoing peritoneal dialysis

DETAILED DESCRIPTION:
Phase I clinical trial which will include ten patients currently undergoing chronic peritoneal dialysis treatment. Patients will be hospitalized for the study. The study will consist of replacing conventional peritoneal dialysis solution with a sodium-free 500 ml solution with 30% icodextrin and 10% dextrose with a dwell time of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients covered by the Mexican Social Security Department.
2. Adults over the age of eighteen.
3. Patients with chronic kidney failure undergoing replacement therapy with peritoneal dialysis.
4. Patients with a functional peritoneal dialysis catheter.
5. Patients undergoing peritoneal dialysis that was stable in the most recent month (ongoing peritoneal dialysis as an outpatient or ongoing cyclic peritoneal dialysis)
6. Patients who wish to participate and who sign the informed consent.
7. If the peritoneal dialysis catheter and the transfer line are compatible with the peritoneal dialysis bag that has a simple luer male connector.
8. If treating doctors consider their patient to be clinically euvolemic.
9. If patients have undergone a peritoneal equilibrium test and their dialysis prescription has not been changed since the test was carried out

Exclusion criteria:

1. Diabetes mellitus type 1 or uncontrolled diabetes (a1c hemoglobin greater than 8%).
2. Active infection.
3. Serum sodium prior to the study less than 130 mmol/l.
4. Serum bicarbonate prior to the study less than 18 mmol/l.
5. Patients who have been prescribed standard peritoneal dialysis who only use solutions with the lowest amount of dextrose
6. Hemoglobin less than 8 g/dl.
7. Active bleeding.
8. Patients prescribed peritoneal dialysis who use a 4.25% dextrose solution at least once a day.
9. Patients with a membrane defect or mechanical defect.
10. Diastolic dysfunction with an increase in filling pressure according to the echocardiogram.
11. Patients with active or suspected peritonitis according to the clinical criterion or their treating doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety defined as the number serious adverse events related to the investigational product | During the 24 hour dwell
  Safety will be described based on the number of serious adverse events that are determined to be related to the investigational product
Tolerability defined as pain in a scale from 0 to 4 during infusion, dwell, and drain | During the 24 hour dwell
  Description of pain. Pain will be described in a scale from 0 to 4; 0 is no pain, 1 is mild pain, 2 is moderate pain, 3 is severe pain, and 4 is extreme pain. Pain will be assessed during infusion, then hourly during the 24 hour dwell, and during the draining

SECONDARY OUTCOMES:
Ultrafiltration | During the 24 hour dwell
  Total volume ultrafiltration as determined by the mL obtained during the draining after the 24hr dwell
Sodium excretion with ultrafiltration | During the 24 hour dwell
  Sodium excretion with ultrafiltration will be calculated by multiplying the mL obtained during the draining after the 24hr dwell by the sodium concentration in a sample of peritoneal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Ivey Miranda, MD, Principal Investigator — Affiliated to Heart Failure Clinic
Locations (1):
- Hospital de Cardiología, Centro Médico Nacional Siglo XXI, Mexico City, Mexico

REFERENCES:
- [Derived] Asher JL, Ivey-Miranda JB, Maulion C, Cox ZL, Borges-Vela JA, Mendoza-Zavala GH, Cigarroa-Lopez JA, Silva-Rueda RI, Revilla-Monsalve C, Moreno-Villagomez J, Ramos-Mastache D, Goedje O, Crosbie I, McIntyre C, Finkelstein F, Turner JM, Testani JM, Rao VS. Development of a Novel Intraperitoneal Icodextrin/Dextrose Solution for Enhanced Sodium Removal. Kidney Med. 2024 Nov 16;7(1):100938. doi: 10.1016/j.xkme.2024.100938. eCollection 2025 Jan. PMID 39790231